CLINICAL TRIAL: NCT00157820
Title: DATAS: The Dual Chamber & Atrial Tachyarrhythmias Adverse Events Study
Acronym: DATAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SP-DATAS
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Results first posted 2012-08-21 (Estimated); Last update posted 2025-07-02 (Actual); Status verified 2024-04

CONDITIONS: Ventricular Tachycardia; Ventricular Fibrillation; Defibrillators, Implantable
Keywords: Defibrillators, Implantable; Atrial Fibrillation; Ventricular Tachyarrhythmias; Clinical Trial
MeSH Terms: conditions — Tachycardia, Ventricular; Ventricular Fibrillation; Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- SC true (Active Comparator): Single chamber Implantable Cardioverter Defibrillator programmed as a Single Chamber.
  Interventions: Device: Single Chamber Implantable Cardioverter Defibrillator
- SC sim (Experimental): Dual chamber ICD initially programmed as single chamber (SC simulated) ICD (''SC sim arm'')
  Interventions: Device: Dual Chamber implantable cardioverter defibrilator
- DC true (Experimental): Dual chamber ICD initially programmed as a DDED (''DC true arm'').
  Interventions: Device: Dual Chamber implantable cardioverter defibrilator

INTERVENTIONS:
Device: Single Chamber Implantable Cardioverter Defibrillator — Single chamber ICD implantation: Medtronic GEM, Medtronic Marquis family of SC ICD
  Other Names: Medtronic GEM, Medtronic Marquis family of SC ICD
  Arms: SC true
Device: Dual Chamber implantable cardioverter defibrilator — Dual chamber ICD implantation: Jewel AF & GemIII AT as DC ICDs (DC true and SC sim arms)
  Other Names: Medtronic Jewel AF, Medtronic GemIII AT, DC ICD
  Arms: DC true; SC sim

SUMMARY:
The Dual Chamber & Atrial Tachyarrhythmias Adverse Events Study (DATAS) was designed to analyze the ability of dual chamber ICDs, to reduce clinically significant adverse events as compared to single chamber ICD in a non selected population with conventional indication of ICD implantation.

DETAILED DESCRIPTION:
Single chamber (SC) implantable cardioverter defibrillators (ICDs) have several limitations that might be relevant during follow up, like atrial pacing requirements, inadequate therapies, sustained atrial tachyarrhythmias and difficulties to achieve an accurate diagnosis of the arrhythmia. Dual chamber (DC) ICDs offer an attractive rationale solution, although controversy remains if the costs and complexity of the implants offer a real clinical advantage.

The DATAS is a, prospective, multicentre, randomized, open labelled study, with three arms (two of them cross-over and the third parallels the other two)

The primary objective of this trial is to determine whether use of Dual Chamber ICD (DDED-DDDR NASPE/BPEG Defibrillator/Pacemaker Codes) results in a significant decrease in the number of primary end points.

The primary end point is a composite comprising four so-denominated "Clinically Significant Adverse Events (CSAE)":

1. all-cause mortality
2. invasive intervention, hospitalization (>24 h) or prolongation of hospitalization due to cardiovascular cause
3. inappropriate shocks (two or more episodes with inappropriate shocks)
4. sustained symptomatic atrial tachyarrhythmias that (a) require urgent termination or (b) last more than 48 h leading to therapeutic intervention.

Secondary objectives are:

1. Number of each of the components of the CSAE.
2. Arrhythmia related: atrial tachyarrhythmia (AT), frequency and burden, ventricular tachyarrhythmia frequency and burden number of appropriate shocks, number of inappropriate shocks, need for reprogramming, need for medication/Radiofrequency Ablation (RFA) for arrhythmia control, pacemaker syndrome and development of dual chamber pacing indication.
3. Cardiovascular related: New York Health Association (NYHA) functional class, exercise capacity, left ventricular ejection fraction (LVEF), reduction of medication (diuretics.).
4. Quality of life: evaluated by the SF-36, Minnesota living test, with heart failure and Symptom Checklist instruments.

ELIGIBILITY:
Inclusion Criteria:

* Meet the Class I implantation criteria for single chamber implantable cardioverter defibrillator according to the guidelines (ACC/AHA).

Exclusion Criteria:

* Permanent atrial fibrillation
* Patients without structural heart disease
* Patient meets implantation criteria for dual-chamber pacing (symptomatic sinus node disease, all 2nd Atrio-Ventricular (AV) block [except asymptomatic Mobitz I] and all 3rd degree AV block ).
* Patient with previous system implanted (ICD or pacemaker).
* Patients with biventricular stimulation or re-synchronization.
* Patient has a mechanical right heart valve.
* Patient has medical conditions that would preclude the testing required by the protocol, or limit study participation.
* Patient is unwilling or unable to cooperate or give written informed consent, or the patient is a minor and legal guardians refuse to give informed consent.
* Patient is or will be inaccessible for follow-up at the study center.
* Patients who are enrolled or planning to enroll in other clinical trials during the clinical study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 354 (Actual)
Dates: Start 2000-11; Primary Completion 2005-05 (Actual); Study Completion 2005-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aurelio Quesada, MD, Principal Investigator — Hospital General Universitario, Valencia, Spain; Jesus Almendral, MD, Principal Investigator — Hospital General Universitario Gregorio Marañon, Madrid, Spain; Fernando Arribas, MD, Principal Investigator — Hospital Universitario 12 de Octubre, Madrid, Spain; Massimo Santini, MD, Principal Investigator — San Filippo Neri Hospital, Rome, Italy; Christian Wolpert, MD, Principal Investigator — University Hospital Mannheim, Mannheim, Germany; Pedro Adragao, MD, Principal Investigator — Santa Cruz Hospital, Carnaxide, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Quesada A, Almendral J, Arribas F, Ricci R, Wolpert C, Adragao P, Cobo E, Navarro X; DATAS Investigators. The DATAS rationale and design: a controlled, randomized trial to assess the clinical benefit of dual chamber (DDED) defibrillator. Europace. 2004 Mar;6(2):142-50. doi: 10.1016/j.eupc.2003.11.011. PMID 15018874
- [Result] Almendral J, Arribas F, Wolpert C, Ricci R, Adragao P, Cobo E, Navarro X, Quesada A; DATAS Steering Committee; DATAS Writing Committee; DATAS Investigators. Dual-chamber defibrillators reduce clinically significant adverse events compared with single-chamber devices: results from the DATAS (Dual chamber and Atrial Tachyarrhythmias Adverse events Study) trial. Europace. 2008 May;10(5):528-35. doi: 10.1093/europace/eun072. Epub 2008 Apr 7. PMID 18390985
- [Result] Ricci RP, Quesada A, Almendral J, Arribas F, Wolpert C, Adragao P, Zoni-Berisso M, Navarro X, DeSanto T, Grammatico A, Santini M; DATAS study Investigators. Dual-chamber implantable cardioverter defibrillators reduce clinical adverse events related to atrial fibrillation when compared with single-chamber defibrillators: a subanalysis of the DATAS trial. Europace. 2009 May;11(5):587-93. doi: 10.1093/europace/eup072. PMID 19401341
- [Result] Hadid C, Almendral J, Ortiz M, Schwab JO, Janko S, Mischke K, Arribas F, Wolpert C, Ricci R, Adragao P, Cobo E, Navarro X, Quesada A. Incidence, determinants, and prognostic implications of true pleomorphism of ventricular tachycardia in patients with implantable cardioverter-defribillators: a substudy of the DATAS Trial. Circ Arrhythm Electrophysiol. 2011 Feb;4(1):33-42. doi: 10.1161/CIRCEP.110.957068. Epub 2010 Nov 13. PMID 21076160

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were eligible if they met a standard Class I indication for a Single Chamber-Implantable Cardioverter Defibrillator (ICD) according to the 1998 ACC/AHA guidelines. Every patient eligible for ICD was screened at each study centre. Follow-up started immediately after randomization.
Pre-assignment Details: The Dual chamber true (DC true) and Single chamber simulated (SC sim) arms crossed over after 8 months. All other crossovers were considered 'premature crossovers' and had to be authorized by an independent Adverse Events Advisory Committee.
  A 1-month wash out period was implemented after programmed crossover.
Groups:
- SC True: Allocated to Single Chamber ICD (SC true arm) VVEV-VVI (NASPE/BPEG Defibrillator/Pacemaker Codes)
- SC Simulated Then DC True: Dual chamber ICD initially programmed as Single Chamber ICD (simulated) then DC true programmed as Dual Chamber true (DDED-DDDR) NASPE/BPEG Defibrillator/Pacemaker Codes.
- DC True Then SC Sim: Dual chamber ICD initially programmed as a DDED-DDDR ("DC true arm") then programmed as Single Chamber simulated
Period: Randomized
Arm/Group | SC True | SC Simulated Then DC True | DC True Then SC Sim
Started | 118 | 116 | 120
Completed | 111 | 111 | 112
Not Completed | 7 | 5 | 8
Not completed — Physician Decision | 4 | 2 | 3
Not completed — Withdrawal by Subject | 1 | 2 | 3
Not completed — Protocol Violation | 2 | 1 | 2
Period: 1st 8 Month
Arm/Group | SC True | SC Simulated Then DC True | DC True Then SC Sim
Started | 111 | 111 | 112
Completed | 103 | 99 | 106
Not Completed | 8 | 12 | 6
Not completed — Death | 7 | 8 | 3
Not completed — Lost to Follow-up | 1 | 2 | 1
Not completed — Premature cross-over | 0 | 2 | 2
Period: 1 Month Wash Out Period
Arm/Group | SC True | SC Simulated Then DC True | DC True Then SC Sim
Started | 103 | 101 (2 patients had crossed over prematurely in SC sim period, that are now carried to DC true period) | 108 (2 patients had crossed over prematurely in DC true period, that are now carried to SC sim period)
Completed | 103 | 101 | 108
Not Completed | 0 | 0 | 0
Period: 2nd 8 Months
Arm/Group | SC True | SC Simulated Then DC True | DC True Then SC Sim
Started | 103 | 101 | 108
Completed | 98 | 88 | 94
Not Completed | 5 | 13 | 14
Not completed — Death | 3 | 1 | 3
Not completed — Lost to Follow-up | 1 | 5 | 2
Not completed — Premature cross-over | 1 | 7 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SC True | SC Simulated Then DC True | DC True Then SC Sim | Total
Number analyzed (Participants) | 111 | 111 | 112 | 334
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 63 | 61 | 53 | 177
  >=65 years | 48 | 50 | 59 | 157
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (10) | 62 (11) | 66 (9) | 64 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 21 | 20 | 52
  Male | 100 | 90 | 92 | 282
Region of Enrollment [Number; unit: participants]
  Spain | 43 | 44 | 44 | 131
  Germany | 29 | 29 | 31 | 89
  Italy | 21 | 21 | 19 | 61
  Israel | 9 | 8 | 9 | 26
  United Kingdom | 6 | 6 | 6 | 18
  Portugal | 3 | 3 | 3 | 9
LVEF [Mean (Standard Deviation); unit: percentage] — Left Ventricle Ejection Fraction (percentage)
  percentage | 35 (13) | 39 (14) | 34 (12) | 36 (13)

OUTCOME MEASURES:

1. Primary Outcome: CSAE-score Rate(Clinical Significant Adverse Events Score Rate)
Description: Main outcome was defined as the CSAE-score during follow-up: CSAE-score rate. We assigned death as the worst outcome during the entire study; and premature cross-over as the main failure of the assigned therapy. So each CSAE was assigned 1 point but (a) death was assigned a score equal to the max number of CSAE in any individual patient in the entire study +1, and (b) premature authorized crossover was given a score equal to the max number of CSAE in any individual patient in that period. Thus, main outcome was defined as the CSAE-score over length of follow-up resulting in a CSAE-score rate.
Time Frame: 17 months
Population: ITT
Measure: Number; unit: score/month
Units Other Than Participants: CSAE
Groups:
- SC True: Allocated to Single Chamber ICD (SC true arm)
- SC Simulated: Dual chamber ICD initially programmed as Single Chamber ICD (simulated)
- DC True: Dual chamber ICD initially programmed as a DDED-DDDR ("DC true arm"
Arm/Group | SC True | SC Simulated | DC True
Number analyzed (Participants) | 111 | 223 | 223
Number analyzed (CSAE) | 82 | 84 | 65
score/month | 0.112 | 0.128 | 0.075
Statistical Analysis 1: Comparison: SC True vs DC True; The assumed effect of the DC treatment was a reduction from 30 to 15% in the proportion of patients who develop a CSAE, as well as a 15% reduction in the mean of CSAE (from 6 to 5.1). The estimated sample size was 200 (DC true) vs. 100 (SC true) patients followed for 8 months, with a two-sided alfa < 0.05 and a power of 88.8%. The sample size was set up to 360 patients (120 patients per arm), considering losses in follow-up; Test type: Superiority or Other; p = 0.0028, Wilcoxon (Mann-Whitney); Odds Ratio (OR) = 0.31, 95% CI 2-sided [0.14 to 0.67] — An additional primary analysis was pre-planned: the odds ratio of CSAE-score between DC and SC obtained from SAS GENMOD procedure with the length of follow-up as an 'offset'

2. Secondary Outcome: Number of Each of the Components of the CSAE
Description: The primary endpoint is a composite of 5 pre-determine Clinical Significant Adverse Events (CSAE): (1) all-cause mortality, (2) invasive intervention due to Cardiovascular cause, (3) hospitalization (>24h) or prolongation of hospitalization due to CV, (4) inappropriate shocks: two or more episodes with inappropriate shocks, (5) sustained symptomatic ATs that (a) require urgent termination or (b) lasted more than 48 h leading to therapeutic intervention.
  Number of each of the components of CSAE, counts the number of events for each pre-determined level.
Time Frame: 17 months
Measure: Number; unit: events
Groups:
- DC True: Dual chamber ICD initially programmed as a DDED-DDDR ("DC true arm")
Arm/Group | SC True | SC Simulated | DC True
Number analyzed (Participants) | 111 | 223 | 223
events
  Death | 10 | 11 | 4
  Invasive intervention CV | 11 | 12 | 10
  Hospitalizations (>24h) or prolongued CV | 42 | 51 | 47
  Inappropiate shocks (>2 episodes) | 13 | 7 | 3
  Long Duration AT | 6 | 3 | 1

ADVERSE EVENTS:
Time Frame: Duration of the enrollment+follow up
Groups:
- SC Simulated: Dual chamber ICD initially programmed as Single Chamber ICD (simulated
Arm/Group | SC True | SC Simulated | DC True
Serious Adverse Events (participants affected / at risk) | 50/111 | 49/223 | 44/223
Other Adverse Events (participants affected / at risk) | 13/111 | 8/223 | 3/223
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SC True (N=111) | SC Simulated (N=223) | DC True (N=223)
Death (General disorders) | 10 (10) | 11 (11) | 4 (4)
Invasive interventions (Cardiac disorders) | 11 (11) | 12 (12) | 9 (10)
Hospitalization or prolongued hospitalizations (Cardiac disorders) | 33 (42) | 32 (51) | 36 (47)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SC True (N=111) | SC Simulated (N=223) | DC True (N=223)
Innapropiate shocks (Cardiac disorders) | 10 (23) | 7 (14) | 2 (5)
Sustain Symptomatic AT (Cardiac disorders) | 5 (6) | 4 (4) | 1 (1) — sustained symptomatic ATs that (a) require urgent termination or (b) lasted more than 48 h leading to therapeutic intervention

LIMITATIONS AND CAVEATS:
The follow-up might have been too short to reveal differences in heart failure-related hospitalizations and related mortality.

Premature crossovers are a limitation of RCT. However, our scoring system severely penalized this cross-overs.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less